CLINICAL TRIAL: NCT06959069
Title: Impact of Intermittent Fasting on Sleep and Quality of Life Among Healthy Adults
Brief Title: Impact of Intermittent Fasting on Sleep and Quality of Life
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Marianna Spinou, Medical Doctor, Université Libre de Bruxelles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: P2024/515/CCB B4062024000365
Record Dates: First submitted 2025-04-17; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Sleep Quality; Quality of Life; Fatigue; Intermittent Fasting
Keywords: intermittent fasting; sleep; quality of life; fatigue
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Fatigue; Intermittent Fasting

STUDY DESIGN:
Intervention Model Description: At recruitment, all subjects will provide their written informed consent prior to enrolling in the study. Once the subject's consent is obtained, the participants will be randomly assigned to Group A or Group B. The study will last 10 weeks in total, with 4 weeks for each intermittent fasting window, followed by a 2-week "washout" period where the subjects follow their usual diet between each group of 4 weeks intermittent fasting period. For the first month, group A will follow a feeding period from 12 p.m. to 8 p.m. (known as late feeding window) and group B will follow a feeding period from 8 a.m. to 4 p.m. (known as early feeding window). The following 2 weeks both groups will return to their usual eating habits (washout period). For the second month, group A will follow an early feeding window while group B will follow a late feeding window.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Fasting - Group A (Active Comparator): Group A will follow intermittent fasting over a feeding period from 12 p.m. to 8 p.m. (known as late feeding window) for one month, then a two weeks period (washout period) that participants will return to their usual eating habits and finally one month of intermittent fasting with a feeding period from 8 a.m. to 4 p.m (early feeding window).
  Interventions: Other: Intermittent Fasting - Late feeding window; Other: Intermittent Fasting - Early feeding window
- Intermittent Fasting - Group B (Active Comparator): Group B will follow intermittent fasting over a feeding period from 8 a.m. to 4 p.m (early feeding window) for one month, then a two weeks period (washout period) that participants will return to their usual eating habits and finally one month of intermittent fasting with a feeding period from 12 p.m. to 8 p.m. (known as late feeding window).
  Interventions: Other: Intermittent Fasting - Late feeding window; Other: Intermittent Fasting - Early feeding window

INTERVENTIONS:
Other: Intermittent Fasting - Late feeding window — Intermittent fasting is an eating pattern that consists of alternating periods of fasting of varying duration with periods of eating. In the present study, all participants will follow a time-restricted feeding/eating (TRF/E) that restricts all dietary intake to an 8- hour daily eating window. There will be two different feeding periods. The first window will allow a feeding period from12 p.m. to 8 p.m. (late feeding window).
Other: Intermittent Fasting - Early feeding window — Intermittent fasting is an eating pattern that consists of alternating periods of fasting of varying duration with periods of eating. In the present study, all participants will follow a time-restricted feeding/eating (TRF/E) that restricts all dietary intake to an 8- hour daily eating window. There will be two different feeding periods. The second window will allow a feeding period from 8 a.m. to 4 p.m (early feeding window).

SUMMARY:
The goal of this clinical trial is to investigate the impact of intermittent fasting on sleep, quality of life and fatigue among healthy volunteers. The main questions aim to answer:

Whether intermittent fasting would allow participants to experience an improvement in their sleep quality, duration and latency? Whether intermittent fasting would ameliorate participants' quality of life and reduce chronic fatigue symptoms? Researchers will compare the two most prevailing fasting windows of intermittent diet including an early morning feeding window (8 a.m.-4 p.m.) and a late feeding window (12 p.m.-8 p.m.) to see if there is a difference among these feeding windows on sleep and quality of life.

Participants will:

* Be divided into two groups (group A and group B) that will alternate their fasting windows.
* Group A will start with intermittent fasting over a feeding period from 12 p.m. to 8 p.m. for one month, then a two weeks period of usual eating habits (washout period) and finally one month of intermittent fasting with a feeding period from 8 a.m. to 4 p.m.
* Group B will follow intermittent fasting over a feeding period from 8 a.m. to 4 p.m for one month, then a two weeks period of usual eating habits (washout period) and finally one month of intermittent fasting with a feeding period from 12 p.m. to 8 p.m.
* At enrollment, at the end of each month of intermittent fasting and at the end of washout period participants will be asked to complete some questionnaires and will be submitted to anthropometric measurements using impedance scales.
* Participants will be asked to complete an electronic 24 hour recall diary using the Automated Self-Administered 24h Dietary Assessment (ASA24) Tool software once per week every week during study.

DETAILED DESCRIPTION:
This is a randomized clinical trial focusing on the effect of intermittent fasting on sleep and quality of life among healthy population. More specifically, the first objective of this study will be to investigate the impact of intermittent fasting on sleep including sleep quality, efficiency, duration, and sleep latency among healthy individuals. The second objective will be to explore the impact of intermittent fasting on participants' quality of life and fatigue using validated questionnaires. The third objective is to compare the effect of the two prevailing fasting windows including early morning feeding window (8 a.m.-4 p.m.) and late feeding window (12 p.m.-8 p.m.) on sleep and quality of life.

The investigators expect that intermittent fasting would have a positive effect on sleep and would allow participants to experience an improvement in their sleep during this practice. The investigators also assume that intermittent fasting would have a positive effect on participants' quality of life and fatigue. Moreover, intermittent fasting during the early morning feeding window (8 a.m.-4 p.m.) would have a more positive impact on sleep and quality of life compared to the late feeding window (12 p.m.-8 p.m.) because it would be more aligned with the circadian rhythm.

This project will be conducted over a 10-week period. Subjects will be divided into two groups (group A and group B) that will alternate their fasting windows each month. Each group will consist of 36 male and female volunteers, adults, aged between 18 and 65 years old, and with a BMI between 18.5 and 29.9.

At recruitment, all subjects will provide their written informed consent prior to enrolling in the study. Once the subject's consent is obtained, the participants will be randomly assigned to Group A or Group B. More specifically, during baseline assessment, the participants will randomly draw an envelope containing a piece of paper labeled Group A or Group B. There will be as many envelopes as there are participants, half containing the Group A paper and the other half containing the Group B paper. Once the subject will be assigned to their group, they will be labeled with a number (ranging from 1 to 36) which will allow us to maintain their anonymity.

The study will last 10 weeks in total, with 4 weeks for each window, followed by a 2-week "washout" period where the subjects follow their usual diet between each group of 4 weeks intermittent fasting period. For the first month, group A will follow a feeding period from 12 p.m. to 8 p.m. (known as late feeding window) and group B will follow a feeding period from 8 a.m. to 4 p.m. (known as early feeding window). The following 2 weeks both groups will return to their usual eating habits. For the second month, group A will follow an early feeding window while group B will follow a late feeding window.

At enrollment, information concerning baseline characteristics such as age, body mass index (BMI), profession, physical activity, usual eating habits and smoking status, will be collected.

During baseline assessment, at the end of each month and at the end of the washout period all participants will complete four validated questionnaires to assess any changes they may have experienced in sleep, quality of life, fatigue, and physical activity. Moreover, during these appointments, anthropometric measurements including height (cm), BMI (kg/m2), muscle mass (kg), visceral mass (kg), fat mass (kg), bone mineral mass (kg), waistline (cm) and waist-hip ratio will be carried out using impedance scales in order to observe any possible changes on body composition. Lastly, participants will be asked verbally to mention if they have experienced any side effects such as headache, vertigo, nausea, vomiting, abdominal pain, changes in bowel movements, fatigue, mood swing.

Subjects will also be required to use the Automated Self-Administered 24h Dietary Assessment (ASA24) Tool software once per week, which is a 24-hour food diary. Its purpose is to collect detailed and accurate information on all foods, beverages, and supplements (vitamins, minerals, etc.) consumed by the subject during the last 24 hours. Data concerning total energy intake (kcal/day), protein intake (gr/day), carbohydrates intake (gr/day), fat intake (gr/day), fibers intake (gr/day), amount of water (L/day) and alcohol intake (gr/day) will be analyzed.

The primary outcome of this study will be to investigate the impact of intermittent fasting on sleep including sleep quality, efficiency, duration, and sleep latency among healthy individuals. This will be carried out using the PSQI - Pittsburgh Sleep Quality Index: a standardized self-report questionnaire assessing the subjective sleep quality, sleep efficiency (percentage of time spent in bed actually asleep), sleep duration, and sleep latency (time taken to fall asleep) over the last month. It consists of 19 items, resulting in a total score of 0 to 21. Scores above 5 can be used as an indicator of poor sleep quality.

The second objective will be to explore the impact of intermittent fasting on participants' quality of life using the validated questionnaire Short Form Health 36 (SF-36) that objectively measures quality of life by covering eight domains of health. Sf-36 assesses eight scales: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, energy/fatigue, social functioning, general mental health (emotional well-being), and role limitations due to emotional health, measured by 36 questions, with an additional question on health change/transition. All scores will be recoded with a maximum score of 100. A higher score indicates a better quality of life.

Another primary outcome that will be explored is the impact of intermittent fasting on symptoms of fatigue. This will be carried out using the Fatigue Assessment Scale (FAS), a 10-item scale assessing symptoms of chronic fatigue.

In addition, the impact of intermittent fasting on physical activity will be examined using the Global Physical Activity Questionnaire (GPAQ). Information concerning participation in physical activity in three areas (work activity, travel to and from places, recreational activities) as well as sedentary behavior will be collecting through 16 questions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects
* Adult subjects - age: between 18 and 65 years old
* Subjects with a BMI between 18.5 and 29.9 kg/m^2
* Male and female subjects

Exclusion Criteria:

* Subjects < 18 years old
* Subjects with Diabetes Mellitus (type 1 and type 2)
* Pregnant and/or breastfeeding and/or postpartum women
* Underweight subjects (BMI < 18.5)
* Obese subjects (BMI > 30)
* Subjects with confirmed sleep disorders (requiring CPAP or sleep medication (sleeping pills))
* Subjects with renal failure (GFR < 30 ml/min/1.73 m^2) or liver disorder
* Subjects with serious cardiovascular, respiratory, neurological, or metabolic medical conditions
* Subjects with malignant tumors
* Subjects with a serious mental disorder requiring medication (e.g., antidepressants or anxiolytics)
* Subjects with eating disorders
* Subjects who have undergone major surgery or have been hospitalized due to major medical condition (surgery, stay in intensive care) within the last one year
* Subjects who have lost more than 10% of their body weight within the last one year
* Subjects actively participating in a weight-loss program
* Subjects with alcohol use disorder (maximum 10 standard alcoholic drinks per week, 2 standard alcoholic drinks per day)
* Subjects with substance use disorder
* Subjects unable to provide informed consent
* Subjects who do not participate simultaneously in another clinical trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Impact of intermittent fasting on sleep | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  The primary outcome of this study will be to investigate the impact of intermittent fasting on sleep including sleep quality, efficiency, duration, and sleep latency among healthy individuals. This will be carried out using the Pittsburgh Sleep Quality Index (PSQI) : a standardized self-report questionnaire assessing the subjective sleep quality, sleep efficiency (percentage of time spent in bed actually asleep), sleep duration, and sleep latency (time taken to fall asleep) over the last month. It consists of 19 items, resulting in a total score of 0 to 21. Scores above 5 can be used as an indicator of poor sleep quality.
Impact of intermittent fasting on quality of life | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  The second objective will be to explore the impact of intermittent fasting on participants' quality of life using the validated questionnaire Short Form Health 36 (SF-36) that objectively measures quality of life by covering eight domains of health. Sf-36 assesses eight scales: physical functioning, role limitations due to physical health, bodily pain, general health perceptions, energy/fatigue, social functioning, general mental health (emotional well-being), and role limitations due to emotional health, measured by 36 questions. All scores are recoded with a maximum score of 100. A higher score indicates a better quality of life.
Impact of intermittent fasting on fatigue | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  Another primary outcome that will be explored is the impact of intermittent fasting on symptoms of fatigue. This will be carried out using the Fatigue Assessment Scale (FAS), a 10-item scale assessing symptoms of chronic fatigue. Each item of the FAS is answered using a 5-point, Likert-type scale ranging from 1 ("never") to 5 ("always"). Total scores range from 10 to 50 with higher scores indicating higher levels of fatigue.

SECONDARY OUTCOMES:
Impact of intermittent fasting on physical activity | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  The impact of intermittent fasting on physical activity will be eamined using the Global Physical Activity Questionnaire (GPAQ). It collects information on physical activity participation in three domains including activity at work, travel to and from places and recreational activities as well as sedentary behaviour, comprising 16 questions.
Effect of intermittent fasting on Body Mass Index | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  Anthropometric measurements including weight in kilograms and height in centimeters will be carried out and combined in order to report Body Mass Index (BMI) in kg/m^2.
Impact of Intermittent fasting on total energy intake | All participants will complete the ASA24 24-hour recall diary once per week for the total 10-week duration of the study (10 times in total). The participants will choose the day during the week that they want to recall their diet.
  Data concerning total energy intake (kilocalories/day) will be analyzed. Subjects will be asked to use the ASA24 (Automated Self-Administered 24h Dietary Assessment Tool) software once per week, which is a 24-hour food diary. Its purpose is to collect detailed and accurate information on all foods, beverages, and supplements (vitamins, minerals, medicinal plants, etc.) consumed by the subject during the last 24 hours.
Effect of intermittent fasting on Muscle Mass | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  Anthropometric measurements including muscle mass estimation in kilograms will be carried out in order to observe any possible changes on body composition.
Effect of intermittent fasting on Visceral Mass | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  Anthropometric measurements including visceral mass estimation in kilograms will be carried out in order to observe any possible changes on body composition.
Effect of intermittent fasting on Fat Mass | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  Anthropometric measurements including fat mass estimation in kilograms will be carried out in order to observe any possible changes on body composition.
Effect of intermittent fasting on Bone Mineral Mass | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  Anthropometric measurements including bone mineral mass estimation in kilograms will be carried out in order to observe any possible changes on body composition.
Effect of intermittent fasting on Waistline | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  Anthropometric measurements including waistline in centimeters will be carried out in order to observe any possible changes on body composition.
Effect of intermittent fasting on Waist-hip Ratio | In total 4 times: at baseline assessment (day 1), at the end of the first month of intermittent fasting (day 28), at the end of the washout period (day 42), at the end of second month of intermittent fasting (day 70)
  Anthropometric measurements including the calculation of waist-hip ratio will be carried out in order to observe any possible changes on body composition.
Impact of Intermittent fasting on Macronutrient intake | All participants will complete the ASA24 24-hour recall diary once per week for the total 10-week duration of the study (10 times in total). The participants will choose the day during the week that they want to recall their diet.
  Data concerning macronutrient intake including protein intake (grams/day), carbohydrates intake (grams/day), fat intake (grams/day) and fibers intake (grams/day) will be analyzed. Subjects will be asked to use the ASA24 (Automated Self-Administered 24h Dietary Assessment Tool) software once per week, which is a 24-hour food diary. Its purpose is to collect detailed and accurate information on all foods, beverages, and supplements (vitamins, minerals, medicinal plants, etc.) consumed by the subject during the last 24 hours.
Impact of Intermittent fasting on water intake | All participants will complete the ASA24 24-hour recall diary once per week for the total 10-week duration of the study (10 times in total). The participants will choose the day during the week that they want to recall their diet.
  Data concerning total amount of water (Liters/day) will be analyzed. Subjects will be asked to use the ASA24 (Automated Self-Administered 24h Dietary Assessment Tool) software once per week, which is a 24-hour food diary. Its purpose is to collect detailed and accurate information on all foods, beverages, and supplements (vitamins, minerals, medicinal plants, etc.) consumed by the subject during the last 24 hours.
Impact of Intermittent fasting on alcohol intake | All participants will complete the ASA24 24-hour recall diary once per week for the total 10-week duration of the study (10 times in total). The participants will choose the day during the week that they want to recall their diet.
  Data concerning alcohol intake (grams/day) will be analyzed. Subjects will be asked to use the ASA24 (Automated Self-Administered 24h Dietary Assessment Tool) software once per week, which is a 24-hour food diary. Its purpose is to collect detailed and accurate information on all foods, beverages, and supplements (vitamins, minerals, medicinal plants, etc.) consumed by the subject during the last 24 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Marianna Arvanitaki, Professor, Study Director — Erasme University Hospital, Gastroenterology Department -Libre University
Locations (1):
- Libre University, Faculty of Human Motor Sciences, Campus Erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
all the individual participant data that uderlie the results reported in this study after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication. No end date.
Access Criteria: researchers who provide a methodologically sound proposal

REFERENCES:
- [Background] Wei X, Cooper A, Lee I, Cernoch CA, Huntoon G, Hodek B, Christian H, Chao AM. Intermittent Energy Restriction for Weight Loss: A Systematic Review of Cardiometabolic, Inflammatory and Appetite Outcomes. Biol Res Nurs. 2022 Jul;24(3):410-428. doi: 10.1177/10998004221078079. Epub 2022 May 8. PMID 35531785
- [Background] Wilkinson MJ, Manoogian ENC, Zadourian A, Lo H, Fakhouri S, Shoghi A, Wang X, Fleischer JG, Navlakha S, Panda S, Taub PR. Ten-Hour Time-Restricted Eating Reduces Weight, Blood Pressure, and Atherogenic Lipids in Patients with Metabolic Syndrome. Cell Metab. 2020 Jan 7;31(1):92-104.e5. doi: 10.1016/j.cmet.2019.11.004. Epub 2019 Dec 5. PMID 31813824
- [Background] Anic K, Schmidt MW, Furtado L, Weidenbach L, Battista MJ, Schmidt M, Schwab R, Brenner W, Ruckes C, Lotz J, Lackner KJ, Hasenburg A, Hasenburg A. Intermittent Fasting-Short- and Long-Term Quality of Life, Fatigue, and Safety in Healthy Volunteers: A Prospective, Clinical Trial. Nutrients. 2022 Oct 10;14(19):4216. doi: 10.3390/nu14194216. PMID 36235868
- [Background] Jensen MD, Ryan DH, Apovian CM, Ard JD, Comuzzie AG, Donato KA, Hu FB, Hubbard VS, Jakicic JM, Kushner RF, Loria CM, Millen BE, Nonas CA, Pi-Sunyer FX, Stevens J, Stevens VJ, Wadden TA, Wolfe BM, Yanovski SZ, Jordan HS, Kendall KA, Lux LJ, Mentor-Marcel R, Morgan LC, Trisolini MG, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines; Obesity Society. 2013 AHA/ACC/TOS guideline for the management of overweight and obesity in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines and The Obesity Society. Circulation. 2014 Jun 24;129(25 Suppl 2):S102-38. doi: 10.1161/01.cir.0000437739.71477.ee. Epub 2013 Nov 12. No abstract available. PMID 24222017
- [Background] Kim BH, Joo Y, Kim MS, Choe HK, Tong Q, Kwon O. Effects of Intermittent Fasting on the Circulating Levels and Circadian Rhythms of Hormones. Endocrinol Metab (Seoul). 2021 Aug;36(4):745-756. doi: 10.3803/EnM.2021.405. Epub 2021 Aug 27. PMID 34474513
- See also: Automated Self-Administered 24-hour (ASA24) Dietary Assessment Tool — https://asa24.nih.gov